CLINICAL TRIAL: NCT05064527
Title: Wrist Angel: A Wearable AI Feedback Tool for OCD Treatment and Research
Brief Title: A Wearable AI Feedback Tool for Pediatric OCD
Status: Completed | Type: Observational
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Technical University of Denmark (Other); University of Copenhagen (Other)
Responsible Party: Sponsor
Other Study IDs: H-18010607- 79689
Record Dates: First submitted 2021-09-07; First posted 2021-10-01 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2022-11

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Signal processing; Oxytocin; Family Accommodation; Biosensor; Mobile app
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva samples will be collected from patients and healthy controls and one of their caregivers at baseline (Week 0) and Week 8 to measure oxytocin concentration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Patients: * OCD (ICD-10 F42) as the primary or secondary diagnosis, verified with a semi-structured psychopathological interview using Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS-PL).
  * CY-BOCS > 7: mild (8-15), moderate (16-23), severe (24-31), extreme (32-40)
  * A psychiatrist determined that the child is eligible for care within psychiatry for their primary diagnosis.
  * Patient is age 8 through 17 years (both inclusive).
  Interventions: Device: wearable biosensor; Behavioral: Treatment as usual (TAU); Behavioral: Exposure and response prevention (ERP)
- Controls: * Ages 8 through 17 years (both inclusive).
  * Sex and age (+/- 3months) matched to an included patient.
  Interventions: Device: wearable biosensor
- Caregivers of Patients: Parent or guardian of patient with OCD
  Interventions: Device: wearable biosensor
- Caregivers of Controls: Parent or guardian of control participant
  Interventions: Device: wearable biosensor

INTERVENTIONS:
Device: wearable biosensor — The E4 wristband will be worn by all groups for the duration of the study. It measures blood volume pulse, electrodermal activity, skin temperature, and movement. Patients will be asked to press the event tagging button when they feel stressed by OCD. Control will be asked to press the button when they feel anxious. Parents will be asked to press the button with they notice their child feels stressed by OCD or anxious.
  Other Names: E4 wristband
Behavioral: Treatment as usual (TAU) — Patients will receive treatment as usual at the child and adolescent mental health center. TAU can range from waitlist to one session of psychoeducation to group or individual psychotherapy to medication.
  Groups: Patients
Behavioral: Exposure and response prevention (ERP) — One ERP session will be offered in Week 0 and Week 8.
  Groups: Patients

SUMMARY:
To test the feasibility of implementing digitally enhanced psychotherapy and research in a community child and adolescent mental health center including the acceptability of the digital technology to patients, parents and therapists.

To use passively collected physiological data and actively collected clinical and biochemical data from the patient and parents to detect and predict episodes of obsessive-compulsive disorder (OCD) -related episodes in children and accommodating behaviour in parents.

DETAILED DESCRIPTION:
Background: Psychiatric and specifically mechanistic research have stagnated mainly due to the time, labour and bias inherent in human-based technologies that dominate the field. To advance translational and precision psychiatry, researchers within psychiatry must forge long-term collaborations with researchers and developers within technology.

Objectives: To improve assessment and psychotherapy for youth obsessive-compulsive disorder (OCD) through developing an artificial intelligence tool to support patients, parents and therapists in cognitive behavioural therapy. To give an innovative push in the public sector hospitals and research through integration of wearable sensors and machine learning techniques.

Methods: 10 patients (8-17 years) and one of their parents from a child and adolescent mental health center will be recruited as in the larger TECTO project. To examine whether the algorithms can distinguish between patients and typically developing children, 10 typically developing sex and age matched children and one of their parents or guardians will also be recruited from the catchment area. Passively sensed physiological indicators of stress are used as input to privacy preserving signal processing and machine learning algorithms, which predict OCD-episodes, clinical severity and family accommodation. Oxytocin, as a biomarker for family accommodation, is measured through saliva samples. Signal processing will be used to extract acoustic and physiological features of importance for therapeutic response.

Expected results: Results from the proposed project will be used to develop artificial intelligence (AI) tools that support clinicians, patients and parents, which will be implemented and evaluated in a public-sector hospital. Technology-enhanced therapy can be used in a stepped care model, in which subclinical symptoms are first monitored using passive sensors and then AI interventions are offered, supported by a healthcare professional, and when outpatient care is needed, the AI tool can support patient engagement. The results of this project will also advance research in computational science and psychiatry by testing biomarkers of clinical relevance.

ELIGIBILITY:
Inclusion Criteria:

* OCD (ICD-10 F42) as the primary or secondary diagnosis, verified with a semi-structured psychopathological interview using K-SADS-PL.
* CY-BOCS > 7: mild (8-15), moderate (16-23), severe (24-31), extreme (32-40)
* A psychiatrist determined that the child is eligible for care within psychiatry for their primary diagnosis.
* Patient is age 8 through 17 years (both inclusive).
* Signed informed consent.

Exclusion Criteria:

* Participation in other OCD trials.
* Comorbid illness that contraindicates trial participation: pervasive developmental disorder not including Asperger's syndrome (ICD-10 F84.0-84.4 + F84.8-84.9)), schizophrenia/paranoid psychosis (ICD-10 F20-25 + F28-29), mania or bipolar disorder (ICD-10 F30 and F31), depressive psychotic disorders (F32.3 + F33.3), substance dependence syndrome (ICD-10 F1x.2).
* Intelligence Quotient <70.
* Any condition (e.g. allergies, eczema, hypersensitivity due to Asperger's syndrome) that would prevent the child or parent from wearing a wristband biosensor.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients: seeking treatment at a child and adolescent mental health center. Controls: living in the catchment area of a the same child and adolescent mental health center.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Binary feasibility | Baseline to Week 8
  Binary feasibility outcomes in terms of recruitment, retention, biosensor functionality, acceptability of the biosensor, adherence to wearing the biosensor, adverse reactions to the biosensor, and physiological, audio, and visual signals as markers of OCD distress, severity and family dynamics. "Success" indicates that the a priori feasibility criteria have been met; "revise" indicates that the criteria have not been met.

OTHER OUTCOMES:
Biosensor experience | Week 7
  Children's and parents' level of physical (dis)comfort of wearing the wristband, degree of satisfaction with the design, concerns of stigmatization and data security as well as usability. There are 13 multiple choice questions answered on a 4-point scale (0 = disagree a lot - 3 = agree a lot ) and one open-ended question.
Wristband compliance | Weeks 0 - 8
  Number of hours parents and children wear the wristband
Adverse reactions - wristband | Weeks 0-8
  Negative effects of the wristband defined as the count of events reported by the parent, child or case worker.
Subjective unit of distress | Week 0 and 8
  Patients rate their level of distress on an 11-point scale (0= no distress; 10 = unbearable distress) during exposure and response prevention sessions.
Symptom hierarchy | Week 0 and 8
  Patients rate their level of distress associated with current OCD symptoms on an 11-point scale (0= no distress; 10 = unbearable distress) on a weekly basis.
Biochemical synchrony | Week 0 and 8
  Correlations between child and parent oxytocin level and response child and parent.
Salivary oxytocin level-child | Weeks 0 and 8
  Concentration of oxytocin in child saliva calculated using Matlab-7 according to relevant standard curves.
Salivary oxytocin level-parent | Weeks 0 and 8
  Concentration of oxytocin in parent saliva calculated using Matlab-7 according to relevant standard curves.
Salivary oxytocin response-parent | Weeks 0 and 8
  Change in oxytocin in parent saliva.
Salivary oxytocin response-child | Weeks 0 and 8
  Change in oxytocin in child saliva.
Family Accommodation Scale - Parent Report (FAS-PR) | Weeks 0, 4, and 8
  Self-rated degree of parental involvement in child OCD symptoms. 13-item measure with 4 subscales: Modifying routines, Participating in rituals, Parental distress caused by accommodating and Child consequences for not accommodating. Parents report the frequency of their accommodating behavior within the past week on 9 items and the severity of stress and consequences on 4 items on a five-point scale (0=never/no to 4= daily/extreme). Total and subscales scores are obtained by summing items.
Family Environment Scale - Parent Report (FES) | Weeks 0
  Self-rated questionnaire in which parents report how they perceive their current family environment. 54 items from the following six subscales are used: 1. Cohesion, 2. Expressiveness, 3. Conflict, 4. Independence, 5. Organization, 6. Control. There are three FES forms (real, ideal, and expectations); only the FES real form will be used, which examines a family member's perception of the family as it is. The scale ranges from 10 to 40, with a score of 10 being representative of no family control and a score of 40 being representative of the greatest magnitude of family control. Therefore, a decrease in score represents a decrease in self-reported family control.
Parental Stress Scale (PSS) | Weeks 0, 4, and 8
  Self-rated degree of stress related to parenting identified child. 18 items rated on 5-point scales. Positively statements are reverse scored. Scores range between 18 and 90. Higher scores reflect greater stress.
KIDSCREEN-52 | Week 0 and Week 8
  Health-related Quality of Life Screening Instrument for Children and Adolescents. Self- and parent-ratings subjective health and well-being on 52 items on 10 subscales. Rasch scores are computed for each dimension (subscale) and are transformed into T-values with a mean of 50 and a standard deviation of 10. Higher scores indicate better quality of life and well-being.
Depression Anxiety Stress Scales (DASS) | Weeks 0
  42-item measure of negative emotional states in adults. Self-rated on a 4-point scale. Scores for Depression, Anxiety and Stress are calculated by summing the scores for the relevant items. Higher scores indicate more depression, anxiety and stress.
Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS) score | Week 0 and Week 8
  Semi-structured clinical interview that measures OCD symptom severity. 10 items, rated from 0 (no symptoms) to 4 (extreme severity), are summed to obtain a total score that can range from 0 to 40. An obsession severity score is obtained by summing the items 1-5. A compulsion severity score is obtained by summing items 6-10.
Clinical Global Impression Severity and Clinical Global Impressions Improvement (CGI-I) | Week 0-8
  Change in severity of psychopathology. At baseline, the one-item CGI-S is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (severely ill). CGI-I scores range from 1 (large improvement) through to 7 (large increase in severity).
OCD symptom remission | Week 0 and Week 8
  30% or more reduction in CY-BOCS score by Week 8. Dichotomous variable.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole N Lønfeldt, PhD, Principal Investigator — Region Capital Denmark; Line Katrine H Clemmensen, PhD, Principal Investigator — Technical University of Denmark; Anne K Pagsberg, MD, PhD, Principal Investigator — Region Capital Denmark
Locations (1):
- Child and Adolescent Mental Health Center - Capital Region of Denmark, Copenhagen, Denmark

REFERENCES:
- [Derived] Olesen KV, Lonfeldt NN, Das S, Pagsberg AK, Clemmensen LKH. Predicting Obsessive-Compulsive Disorder Events in Children and Adolescents in the Wild using a Wearable Biosensor (Wrist Angel): Protocol for the Analysis Plan of a Nonrandomized Pilot Study. JMIR Res Protoc. 2023 Nov 14;12:e48571. doi: 10.2196/48571. PMID 37962931
- [Derived] Lonfeldt NN, Olesen KV, Das S, Mora-Jensen AC, Pagsberg AK, Clemmensen LKH. Predicting obsessive-compulsive disorder episodes in adolescents using a wearable biosensor-A wrist angel feasibility study. Front Psychiatry. 2023 Oct 2;14:1231024. doi: 10.3389/fpsyt.2023.1231024. eCollection 2023. PMID 37850105
- [Derived] Lonfeldt NN, Clemmensen LKH, Pagsberg AK. A Wearable Artificial Intelligence Feedback Tool (Wrist Angel) for Treatment and Research of Obsessive Compulsive Disorder: Protocol for a Nonrandomized Pilot Study. JMIR Res Protoc. 2023 Jul 24;12:e45123. doi: 10.2196/45123. PMID 37486738